CLINICAL TRIAL: NCT00913744
Title: A Randomized, Sham-Injection Controlled, Double-Masked, Multicenter Trial of Ocriplasmin Intravitreal Injection for Treatment of Focal Vitreomacular Adhesion in Subjects With Exudative Age-Related Macular Degeneration (AMD)
Brief Title: Safety and Efficacy Study of Intravitreal Ocriplasmin in Subjects With AMD With Focal Vitreomacular Adhesion
Acronym: MIVI-5
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ThromboGenics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TG-MV-005
Record Dates: First submitted 2009-06-02; First posted 2009-06-04 (Estimated); Results first posted 2014-05-05 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-04

CONDITIONS: Exudative Age-Related Macular Degeneration; Focal Vitreomacular Adhesion
Keywords: AMD
MeSH Terms: interventions — microplasmin; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ocriplasmin (Experimental)
  Interventions: Drug: Ocriplasmin
- Sham injection (Sham Comparator)
  Interventions: Drug: Sham injection

INTERVENTIONS:
Drug: Ocriplasmin — ocriplasmin intravitreal injection (125 µg)
  Arms: Ocriplasmin
Drug: Sham injection — Sham injection
  Arms: Sham injection

SUMMARY:
This study will evaluate the safety and efficacy of Ocriplasmin intravitreal injection, in subjects diagnosed with exudative AMD with focal vitreomacular adhesion. Ultimately, it is believed that intravitreal ocriplasmin may offer physicians a safe agent for pharmacologic vitreolysis and nonsurgical resolution of focal vitreomacular adhesion in AMD subjects where this adhesion may be causally associated with worse prognosis).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged > 50
2. Presence of focal vitreomacular adhesion measured by Optical Coherence Tomography (OCT).
3. Diagnosis of active primary or recurrent subfoveal CNV secondary to AMD, including those with predominantly classic, minimally classic or occult lesions with no classic component.
4. The total area of Choroidal Neovascularization (CNV) (including both classic and occult components) encompassed within the lesion must be > 50% of the total lesion area
5. The total lesion area must be < 12 disc areas
6. Subjects who have previously received at least three antiangiogenic injections(Lucentis® or Avastin®) in the study eye.
7. Subjects with visual acuity of 20/32 to 20/200 in the study eye
8. Written informed consent obtained from the subject prior to inclusion in the study

Exclusion Criteria:

1. Evidence of complete macular Posterior Vitreous Detachment (PVD) in the study eye on biomicroscopy, B-scan ultrasound or OCT prior to planned study drug injection
2. Subjects with vitreous haemorrhage which precludes either of the following: visualization of the posterior pole by visual inspection or adequate assessment of the macula by either OCT and/or fluorescein angiography in the study eye or other opacities precluding visualisation of the fundus.
3. Subjects who have previously received more than 9 antiangiogenic agent injections (whether Lucentis® or Avastin® or other anti-angiogenic agent) in the study eye
4. Subjects with history of rhegmatogenous retinal detachment or proliferative vitreoretinopathy (PVR) in the study eye
5. Subjects with high myopia (> 8D) or aphakia in the study eye
6. Subjects who have had ocular surgery in the study eye in the prior three months
7. Subjects who have had a vitrectomy in the study eye at any time.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-01; Primary Completion 2012-12 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (27):
- United States (12):
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Retinal Consultants Medical Group, Sacramento, California
  - University of Colorado Denver, Aurora, Colorado
  - Center for Retina and Maculla Disease, Winter Haven, Florida
  - Southeast Retina Center, PC, Augusta, Georgia
  - VitreoRetinal Surgery, PA, Minneapolis, Minnesota
  - Retina-Vitreous Center, PA, New Brunswick, New Jersey
  - Allegheny Ophthalmic & Orbital Associates, PC, Pittsburgh, Pennsylvania
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Southeastern Retina Associates, Kingsport, Tennessee
  - Retinal Consultants of Houston,, Houston, Texas
  - Valley Retina Institute, McAllen, Texas
- U.Z. Leuven St. Rafaël Hospital, Leuven, Belgium
- France (4):
  - Rabelais Ophthalmologic Center, Lyon
  - Centre Paradis-Monticelli, Marseille
  - Centre Ophtalmologique d'Imagerie et de Laser, Paris
  - Centre Ophtalmologique de L'Odeon, Paris
- Germany (4):
  - Universität Bonn Augenklinik, Bonn
  - Universität Lübeck Universitätsklinikum Schleswig-Holstein, Lübeck
  - Klinik für Augenheilkunde, Universitätsklinikum Gießen, Standort Marburg, Marburg
  - Augenklinik der Ludwig Maximilians Universität München, München
- Italy (2):
  - University of Milan Department of Clinical Science "Luigi Sacco", Milan
  - Largo Agostino Gemelli (University Hospital) Institute of Ophthalmology, Rome
- United Kingdom (4):
  - Frimley Park Hospital, Frimley, Camberley
  - Royal Liverpool & Broadgreen Hospital, Liverpool
  - Moorfields Eye Hospital, London
  - Wolverhampton Eye Infirmary New Cross Hospital, Wolverhampton

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject was enrolled on 29 Jan 2010 and last subject completed the study on 06 Dec 2012
Groups:
- Ocriplasmin: Intravitreal injection (125 µg)
- Sham: Sham injection
Period: Overall Study
Arm/Group | Ocriplasmin | Sham
Started | 75 | 25
Completed | 70 | 24
Not Completed | 5 | 1
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): All randomized subjects who have been administered trial medication and for whom data of at least one post-baseline efficacy assessment is available. One subject (ocriplasmin) was not included in the FAS because the subject withdrew consent after receiving study treatment and refused further contact.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ocriplasmin | Sham | Total
Number analyzed (Participants) | 74 | 25 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.5 (8.13) | 74.7 (7.16) | 74.6 (7.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 15 | 54
  Male | 35 | 10 | 45

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With Focal Vitreomacular Adhesion (VMA) Release by Day 28
Description: The VMA release was determined by masked Central Reading Center Optical Coherence Tomography (OCT) evaluation
Time Frame: Day 28
Population: The Full Analysis Set (FAS) was the primary data set for efficacy analysis. Data that were missing for any reason were imputed using the Last Observation Carried Forward (LOCF) method.
Measure: Number; unit: percentage of subjects
Arm/Group | Ocriplasmin | Sham
Number analyzed (Participants) | 74 | 25
percentage of subjects | 24.3 | 12.0
Statistical Analysis 1: Comparison: Ocriplasmin vs Sham; Test type: Superiority or Other; p = 0.262, Fisher Exact; P-value is from Fisher's exact test, comparing sham and ocriplasmin; Difference in proportions = 12.3, 95% CI 2-sided [-3.7 to 28.4]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs)/Serious Adverse Events (SAEs) were collected from injection day up to discontinuation, and for a maximum of 12 months after injection.
Description: Safety Set consisted of all subjects who received study treatment and was used for all safety analysis. All subjects were included in the Safety Set: 75 subjects in the ocriplasmin group and 25 subjects in the sham group. AEs and SAEs include ocular events in study eye and non-study eye, as well as non-ocular events.
Arm/Group | Ocriplasmin | Sham
Serious Adverse Events (participants affected / at risk) | 18/75 | 2/25
Other Adverse Events (participants affected / at risk) | 33/75 | 11/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ocriplasmin (N=75) | Sham (N=25)
Retinal detachment (Eye disorders) | 3 (3) | 0 (0)
Visual acuity reduced (Eye disorders) | 3 (3) | 0 (0)
Blindness transient (Eye disorders) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Endophthalmitis (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Vocal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Intraocular pressure increased (Investigations) | 2 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1)
Vocal cordectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Ateriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ocriplasmin (N=75) | Sham (N=25)
Visual acuity reduced (Eye disorders) | 12 (17) | 3 (5)
Photopsia (Eye disorders) | 9 (10) | 2 (2)
Eye pain (Eye disorders) | 10 (10) | 0 (0)
Conjuctival haemorrhage (Eye disorders) | 7 (8) | 2 (3)
Retinal haemorrhage (Eye disorders) | 3 (3) | 5 (6)
Vitreous floaters (Eye disorders) | 8 (9) | 0 (0)
Blepharitis (Eye disorders) | 4 (4) | 0 (0)
Cataract nuclear (Eye disorders) | 4 (4) | 0 (0)
Corneal oedema (Eye disorders) | 4 (4) | 0 (0)
Metamorphosia (Eye disorders) | 1 (1) | 2 (2)
Ulcerative keratitis (Eye disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and the Principal Investigator (PI) reserve the right to publish only the results of the work performed by the Principal Investigator pursuant to this Agreement; provided, however, that Institution provides Sponsor a copy of any proposed publication, for review and comment at least sixty (60) days in advance of its submission for publication.